CLINICAL TRIAL: NCT02947035
Title: Molecular Testing to Direct Extent of Initial Thyroid Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Linwah Yip, MD, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19050280
Record Dates: First submitted 2016-10-20; First posted 2016-10-27 (Estimated); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; thyroid nodule; thyroidectomy; personalized medicine
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule | interventions — Cyclin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Risk (Experimental): Molecular testing and ultrasound features will be used to predict if thyroid cancer is low risk. Intervention will be to perform thyroid lobectomy.
  Interventions: Procedure: Thyroid lobectomy
- High Risk (Experimental): Molecular testing and ultrasound features will be used to predict if thyroid cancer is high risk. Intervention will be to perform more aggressive surgery to include total thyroidectomy with CCND.
  Interventions: Procedure: Total thyroidectomy with CCND

INTERVENTIONS:
Procedure: Thyroid lobectomy — Thyroid lobectomy is removal of only part of the thyroid
  Arms: Low Risk
Procedure: Total thyroidectomy with CCND — Total thyroidectomy with central compartment lymph node dissection is removal of the entire thyroid with the surrounding lymph nodes
  Arms: High Risk

SUMMARY:
The research study consists of the participant agreeing to 1) the use of preoperative molecular testing (ThyroSeq) to guide extent of initial surgery and 2) the prospective collection of medical record data related to treatment of thyroid cancer.

DETAILED DESCRIPTION:
The aim of the proposed pilot study is to use a clinical algorithm that incorporates molecular, clinical and radiographic factors to inform surgical management. This study is the first to propose molecular-directed surgical management for this commonly diagnosed cancer.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid nodule is >1.5 cm
* Preoperative FNA biopsy that is positive for papillary thyroid cancer or suspicious for papillary thyroid cancer

Exclusion Criteria:

* Prior thyroid/parathyroid surgery
* Clinical indications for total thyroidectomy including hypothyroidism, history of head or neck radiation when <18 years old
* Recurrent laryngeal nerve dysfunction
* Diagnosis of concurrent primary hyperparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who require completion thyroidectomy for aggressive histology features | 2 years
  Histology characteristics of tumor will be assessed including type of cancer, extrathyroidal extension, lymph node metastasis, and margin status to assess if completion thyroidectomy is needed per the 2015 ATA guidelines

SECONDARY OUTCOMES:
Number of patients who had central compartment neck dissection but no lymph node metastasis were identified | 2 years
Number of patients with operative complications | 2 years
  incidence of permanent nerve injury, hypocalcemia, readmission
Recurrence | >2 years
QOL metric - FACT-G cumulative score preop, postop, and at followup | 2 years
QOL metric - QOL-Thyroid cumulative score preop, postop, and at followup | 2 years
QOL metric - SF36 cumulative score preop, postop, and at followup | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Linwah Yip, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No